CLINICAL TRIAL: NCT03794856
Title: The Dallas Asthma Brain and Cognition (ABC) Study
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Sherwood Brown, MD, PhD, Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU-2018-0034
Record Dates: First submitted 2018-12-12; First posted 2019-01-07 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Asthma
Keywords: Healthy participants; Asthma; Cognitive functioning; MRI
MeSH Terms: conditions — Asthma | interventions — Functional Status

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Asthma patients: Asthma patients will undergo behavioral testing and imaging at a single timepoint.
  Interventions: Other: Functional and Structural Magnetic Resonance Imaging (research grade); Other: Cognitive Function Testing (non-diagnostic); Other: Asthma and Psychological Questionnaires (non-diagnostic)
- Healthy Volunteers: Healthy volunteers will undergo behavioral testing and imaging at a single timepoint.
  Interventions: Other: Functional and Structural Magnetic Resonance Imaging (research grade); Other: Cognitive Function Testing (non-diagnostic); Other: Asthma and Psychological Questionnaires (non-diagnostic)

INTERVENTIONS:
Other: Functional and Structural Magnetic Resonance Imaging (research grade) — Brain structure and function will be compared in middle to late-age adults with asthma compared to healthy adults.
Other: Cognitive Function Testing (non-diagnostic) — Multiple domains of cognitive functioning will be investigated, including processing speed, executive functioning/working memory and episodic memory.
Other: Asthma and Psychological Questionnaires (non-diagnostic) — Participants will fill out asthma and psychological questionnaires (non-diagnostic)

SUMMARY:
Asthma is a chronic inflammatory airway disease that leads to episodic symptom exacerbations, which exerts a substantial burden on quality of life and can influence other health domains if not adequately controlled. Asthma prevalence rates have increased in the past decade, affecting 8.4% (25.7 million people) of the United States population. The economic costs of asthma have been estimated annually with $56 billion in the US alone. Despite progress in pharmacological treatment, overall asthma control remains unsatisfactory and treatment non-adherence is extremely high. Asthma is particularly under diagnosed and understudied in aging adults. This problem will increase in coming decades given demographic trends and will disproportionally contribute to the societal and personal economic costs associated with asthma treatment and management. In the proposed 4-year project we will evaluate, in a two-session assessment recruiting a total of 126 asthma patients and 66 healthy controls aged 40-69 years, the extent to which asthma and aging are associated with changes in cognition and brain chemistry, structure, and function.

DETAILED DESCRIPTION:
This study will implement a cross-sectional design, conducted across two sessions. The first session will capture cognitive performance, health history, and relevant social, behavioral, and emotional processes. The second session approximately one week later will capture neural structure, function, and chemistry. In the first session, participants will undergo screening for psychological disorders, neuropsychological testing and pulmonary function assessment at the Southern Methodist University (SMU) or UT Southwestern site. They will then participate in a second session at University of Texas Southwestern Medical Center (UTSW) Advanced Imaging Research Center (AIRC) with structural and functional magnetic resonance imaging (MRI), diffusion tensor imaging (DTI), and brain metabolic activity with spectroscopy. Blood draws and additional pre- and post-neuroimaging spirometry will also be performed at the second session. Potential participants identified by brief phone screen will be invited for two assessment sessions 1 week apart. At the first session, they will be consented, interviewed about their asthma and/or general health status, and pulmonary function tests will be performed. They will then fill in questionnaires and will be screened for psychological disorders by standardized psychiatric interview. After that, they will complete the neuropsychological test battery. The second session will entail spirometry (to ascertain adequate lung function for imaging), the 1 ½ hour neuroimaging protocol, saliva samples, and blood sampling. Spirometry will be repeated at the end of the imaging session. We will also offer patients a brief optional session before the imaging session to get acquainted to the scanning environment in a mock scanner.

ELIGIBILITY:
Inclusion Criteria:

* For asthma patients: diagnosis of asthma (verified by a medical documentation) for at least 2 years; for healthy volunteers: no significant medical or psychiatric history.
* Ages 40 to 69 years old.
* Proficient in English.
* Education level of at least 10th grade level.

Exclusion Criteria:

* Treatment with oral corticosteroids in the previous 6 weeks, because of the potent effects of this drug on airway reactivity.
* Spirometry: Peak expiratory flow (PEF) below 60% of predicted.
* Diagnosis of vocal cord dysfunction (identified by abnormalities in spirometric flow-volume curves), clinically significant chronic obstructive pulmonary disease, or emphysema.
* Presence or history of medical or neurological disorder that may affect brain function and the physiological systems of interest (e.g. angina, myocardial infarction, congestive heart failure, transient ischemic attacks, cerebrovascular accidents, emphysema, or chronic obstructive pulmonary disease, history of seizures or head trauma, endocrine disorders or renal disease, chemotherapy or radiation presently or in the past 5 years, uncontrolled diabetes, blood pressure above 160/90 (self-reported or measured at session 1).
* Corrected vision poorer than 20/30 on Snellen Eye Chart.
* Presence or history of Schizophrenia, Psychosis, Dementia, Bipolar I, Bipolar II, PTSD or Acute Stress Disorder
* Current or recent history (within 1 year) of Substance Related Disorders, current recreational drug use (defined as past 30 days) or consuming more than 20 alcoholic drinks per week.
* Current treatment with anti-psychotics, sedatives, benzodiazepines with a half-life longer than 6 hours.
* Previous electroconvulsive therapy.
* Presence of history of orthopaedic circumstances and metallic inserts interfering with MR scanning (prior surgeries and/or implant pacemakers, pacemaker wires, artificial heart value, brain aneurysm surgery, middle ear implant, non-removable hearing aid or jewelry, braces or extensive dental work, cataract surgery or lens implant, implanted mechanical or electrical device, artificial limb or joint, foreign metallic objects in the body such as bullets, BB's, shrapnel, or metalwork fragments, pregnancy, claustrophobia, uncontrollable shaking, or inability to lie still for one hour.
* Not proficient in English.
* In the opinion of the principal investigator, participant is otherwise unsuitable for this study.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the larger Dallas/ Fort Worth community. We will recruit both healthy controls and subjects with asthma through local flyers, online advertisements, at community allergy and pulmonary clinics, and databases. Individuals who appear eligible will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Examine processing speed of middle- to late-age adults with asthma with the Wechsler Adult Intelligence Scale (WAIS) Symbol Search Test. | From date of baseline until the date of second session, approximately one week after baseline.
  The Wechsler Adult Intelligence Scale (WAIS) Symbol Search test is a subtest of the WAIS, a scale widely used to measure intelligence. The examinee scans a search group of symbols and indicates whether one of the symbols matches a symbol in the target group. The time limit for this subtest is 120 seconds. The total raw score is the sum of the number of correct responses minus the number of incorrect responses. A higher score indicates better performance. The maximum total raw score is 60. If the total raw score is equal to or less than 0, then the total raw score is recorded as 0.
Examine executive functioning of middle- to late-age adults with asthma with the Trails A&B test. | From date of baseline until the date of second session, approximately one week after baseline.
  The Trails A&B test is a neuropsychological assessment. The task requires a subject to connect a sequence of 25 circles on a sheet of paper as quickly as possible. The test has 2 parts, with the first part of the test requiring the subject to connect circles that are all numbers (1, 2, 3, etc.) in order. The second part of the test requires that the subject alternates between numbers and letters (1, A, 2, B, etc.). The time taken for each part, measured in seconds, is the raw score. The score is then converted to a scaled score and a T score, both based on sex (male, female), race, and age. A higher score indicates better performance.
Examine working memory of middle- to late-age adults with asthma with the National Institute of Health (NIH) Sorting Working Memory Test. | From date of baseline until the date of second session, approximately one week after baseline.
  The National Institute of Health Sorting Working Memory Test is a computerized test that requires the subject to sequence sets of visually and auditorily presented stimuli (pictures of animals and food) in size order from smallest to biggest. There are two lists, with the 1-list version requiring sequencing among a single category (either animals or food), and the 2-list version (requiring sequencing of both food and animals within a series). The raw score is based on the sum of the correct across both lists, which comprise the List Sorting "Total Score". The raw score is converted into a t-score (mean = 50, standard deviation = 10). A higher score indicates better performance.
Examine episodic memory of middle- to late-age adults with asthma with the Rey Auditory Verbal Learning Test (RAVLT). | From date of baseline until the date of second session, approximately one week after baseline.
  The examiner reads a list of 15 nouns aloud at the rate of one per second. The subject is asked to repeat all words they recall over 5 trials. An interference list (List B) is then read and subject is asked to recall. Immediately following the interference trial, the subject is asked to recall words from List A (Trial 6). After a 20 minute delay the subject is asked to recall as many words as possible from the first list (delayed recall). A list of 50 words is presented containing all words from List A and the subject is asked to indicate whether each word was on List A (recognition task). The total score (Trials 1-5) is calculated by summing the correct number of words for each trial. List B, Trial 6 and Delayed Recall are calculated by summing the correct number of words. Recognition task is scored by taking the number of correct words and subtracting the number of false positive words. Scores are converted into t-scores with higher score indicating better performance.
Examine reasoning of middle- to late-age adults with asthma with the National Adult Reading Test (NART). | From date of baseline until the date of second session, approximately one week after baseline.
  The National Adult Reading Test is a commonly used test to measure intellectual ability in English-speaking patients. A list of 50 words, whose pronunciation cannot be determined from their spelling, are given to the subject and the subject is asked to read down the list. The examiner marks whether the subject pronounced the word correctly and the NART is scored by summing the number of words pronounced correctly.
Examine brain function of adult asthma patients from age 40-69 with functional magnetic resonance imaging (fMRI) | From date of baseline until the date of second session, approximately one week after baseline.
  We will assess brain functioning by measuring default brain network connectivity using functional magnetic resonance imaging (fMRI)
Examine brain structure of adult asthma patients from age 40-69 with structural magnetic resonance imaging (sMRI) | From date of baseline until the date of second session, approximately one week after baseline.
  We will assess brain structure, hippocampal gray matter volume, using structural magnetic resonance imaging (sMRI)
Examine brain chemistry of adult asthma patients from age 40-69 with proton magnetic resonance spectroscopy (1H-MRS) | From date of baseline until the date of second session, approximately one week after baseline.
  We will assess brain chemistry, specifically differences in hippocampal metabolite levels, using proton magnetic resonance spectroscopy (1H-MRS)

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Southern Methodist University, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No